CLINICAL TRIAL: NCT03595163
Title: Effects of Propofol and Sevoflurane on Blood Folic Acid and Homocysteine Concentrations in Children With Cochlear Implant Surgery
Brief Title: Effects of Propofol and Sevoflurane on Blood Folic Acid and Homocysteine Concentrations in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Jingjie Li, vice-director, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2018-121-T99
Record Dates: First submitted 2018-07-02; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Sevoflurane; Propofol; Homocysteine; Cochlear Hearing Loss
Keywords: Sevoflurane; Propofol; Folic Acid Concentrations; Homocysteine Concentrations; Cochlear Implant Surgery
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Experimental): Children aged 1 month to 3 years who were scheduled to undergo cochlear implant surgery under general anesthesia were enrolled in this study.Children were treated with an infusion bolus of 2.0mg/kg propofol during anesthesia induction and maintained with 2.0-2.5vol% sevoflurane, with the dosage adjusted to achieve loss of consciousness.The bispectral index of EEG was maintained between 50 and 60 in all groups.The homocysteine and folic acid concentrations were measured after anesthesia induction and at the end of surgery separately .
  Interventions: Drug: Sevoflurane
- Group P (Active Comparator): Children aged 1 month to 3 years who were scheduled to undergo cochlear implant surgery under general anesthesia were enrolled in this study.Children were treated with an infusion bolus of 2.0mg/kg propofol during anesthesia induction and continuous infusion of 7 to 8mg/kg/hour, with the dosage adjusted to achieve loss of consciousness.The bispectral index of EEG was maintained between 50 and 60 in all groups.The homocysteine and folic acid concentrations were measured after anesthesia induction and at the end of surgery separately .
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — After anesthesia induction and at the end of the operation, all patients were taken 2-3ml arterial blood respectively.The blood was put at normal temperature for 30 minutes.Then the serum was centrifuged to measure the homocysteine and folic acid concentrations.
  Other Names: Blood Folic Acid and Homocysteine Concentrations
  Arms: Group S
Drug: Propofol — After anesthesia induction and at the end of the operation, all patients were taken 2-3ml arterial blood respectively.The blood was put at normal temperature for 30 minutes.Then the serum was centrifuged to measure the homocysteine and folic acid concentrations.
  Other Names: Blood Folic Acid and Homocysteine Concentrations
  Arms: Group P

SUMMARY:
To investigate the effect of sevoflurane and propofol on the concentrations of serum homocysteine and folic acid in children who received cochlear implant surgery.

DETAILED DESCRIPTION:
This study is a prospective single center, cross-reference clinical application study.This study plan to enroll 40 children with cochlear implant surgery. Children were selected randomly and divided into 2 groups.Each group has 20 patients. All children undergo orotracheal intubation, mechanical ventilation will given by anaesthetic machine (U.S. Ohmeda advance cs2 ) to maintain oxygen saturation above 95%, hemodynamics and other vital signs were monitored with the anesthesia monitor.In the operation room,2-3ml arterial blood will be taken.And the levels of homocysteine and folic acid will be measured at week 1.

ELIGIBILITY:
Inclusion Criteria:

* children accepted cochlear implant surgery under general anesthesia
* no participate in any other trial up to 3 months before this study
* no acute infectious diseases, systemic diseases
* willing to participate in this study and sign the informed consent

Exclusion Criteria:

* unwilling to participate in this study
* with a history of serious liver or kidney dysfunction
* hemodynamic instability (etc. shock, blood pressure reduced by 30%)
* children with egg milk allergy
* children with a family history of malignant hyperthermia

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Serum folate levels | Measured at Week 1
  The serum folate concentration was detected by microparticle enzyme immunoassay.

SECONDARY OUTCOMES:
Plasma homocysteine levels | Measured at Week 1
  The serum homocysteine concentration was detected by fluorescence polarization immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Hong, Ph.D, Study Director — Shanghai9 hospital; Li Jingjie, Ph.D, Study Chair — Shanghai9 hospital
Locations (1):
- Shanghai ninth people's hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez-Vega R, Garrido F, Partearroyo T, Cediel R, Zeisel SH, Martinez-Alvarez C, Varela-Moreiras G, Varela-Nieto I, Pajares MA. Folic acid deficiency induces premature hearing loss through mechanisms involving cochlear oxidative stress and impairment of homocysteine metabolism. FASEB J. 2015 Feb;29(2):418-32. doi: 10.1096/fj.14-259283. Epub 2014 Nov 10. PMID 25384423
- [Background] Cadoni G, Agostino S, Scipione S, Galli J. Low serum folate levels: a risk factor for sudden sensorineural hearing loss? Acta Otolaryngol. 2004 Jun;124(5):608-11. doi: 10.1080/00016480410016216. PMID 15267180
- [Background] Krapels IP, Vermeij-Keers C, Muller M, de Klein A, Steegers-Theunissen RP. Nutrition and genes in the development of orofacial clefting. Nutr Rev. 2006 Jun;64(6):280-8. doi: 10.1111/j.1753-4887.2006.tb00211.x. PMID 16808114
- [Background] Verkleij-Hagoort A, Bliek J, Sayed-Tabatabaei F, Ursem N, Steegers E, Steegers-Theunissen R. Hyperhomocysteinemia and MTHFR polymorphisms in association with orofacial clefts and congenital heart defects: a meta-analysis. Am J Med Genet A. 2007 May 1;143A(9):952-60. doi: 10.1002/ajmg.a.31684. PMID 17431894
- [Background] Coskunfirat N, Hadimioglu N, Ertug Z, Akbas H, Davran F, Ozdemir B, Aktas Samur A, Arici G. Homocysteine levels after nitrous oxide anesthesia for living-related donor renal transplantation: a randomized, controlled, double-blind study. Transplant Proc. 2015 Mar;47(2):313-8. doi: 10.1016/j.transproceed.2014.10.014. Epub 2015 Jan 31. PMID 25648379
- See also: Methylene Tetrahydrofolate Reductase Deficiency: the Hidden Risk in Paediatric Anaesthesia. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Methylene+Tetrahydrofolate+Reductase+Deficiency%3A+the+Hidden+Risk+in+Paediatric+Anaesthesia.+Turk+J+Anaesthesiol+Reanim